CLINICAL TRIAL: NCT05206266
Title: Bioenhancing Effects of Black Pepper With Turmeric on Pain Ratings: a Randomized, Clinical Trial
Brief Title: Bioenhancing Effects of Black Pepper With Turmeric on Pain Ratings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Principal Investigator, Daniel L. Smith, Jr., Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300005070
Record Dates: First submitted 2021-12-13; First posted 2022-01-25 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turmeric, then Turmeric+Black Pepper (Experimental): Participants first receive Turmeric (Turmeric provided at 300mg, 1g or 3g; n=10 subjects/amount with no black pepper) for 1 week. After a 1 week washout, participants then receive Turmeric at the previous amount plus Black Pepper (Turmeric provided at 300mg, 1g or 3g daily; n=10 subjects/amount and Black Pepper 300mg/subject daily) for 1 week.
  Interventions: Other: Turmeric; Other: Turmeric+Black Pepper
- Turmeric+Black Pepper, then Turmeric (Experimental): Participants first receive Turmeric+Black Pepper (Turmeric provided at 300mg, 1g or 3g daily; n=10 subjects/amount and Black Pepper at 300mg/subject daily) for 1 week. After a 1 week washout, participants then receive Turmeric daily at the previous amount for 1 week (Turmeric provided at 300mg, 1g or 3g; n=10 subjects/amount with no black pepper).
  Interventions: Other: Turmeric; Other: Turmeric+Black Pepper

INTERVENTIONS:
Other: Turmeric — Three amounts of dietary turmeric will be tested: 1) turmeric 300 mg/day, 2) turmeric 1 g/day, 3) turmeric 3 g/day.
Other: Turmeric+Black Pepper — Three amounts of dietary turmeric (300mg/day, 1g/day or 3g/day) with black pepper (300 mg) added to the turmeric.

SUMMARY:
Although multiple clinical trials have been reported studying the effects of turmeric and turmeric-derived curcuminoid containing extract on pain by various study designs (including both acute and chronic pain), with the most consistent positive pain reduction benefits at turmeric or curcuminoid levels above normal dietary intake estimates, studies assessing the combination of black pepper and turmeric at culinary relevant levels for pain remediation benefits are needed. As black pepper is reported to 'enhance' the effects of co-consumed compounds, we are testing whether consumption of black pepper alters the pain alleviating effects of turmeric when consumed at levels representative of potential dietary intakes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 or older
* BMI: 20-40
* Diet: No dietary prohibitions/allergies
* 21-day availability
* Moderate Pain Rating (self-reported numeric rating 4-7 on 10 pt scale)

Exclusion Criteria:

* Turmeric or Black Pepper Allergy, or any allergy that would prevent menu item selections for 7 days of feeding
* Recent change in pain levels - e.g. acute injury
* Known eating disorder
* No access to a phone capable of text message, electronic device (phone, tablet, computer/laptop) with email and internet access
* Inability to continue on protocol for 3 consecutive weeks.
* Medical conditions (cardiovascular disease event within the past six months, severe pulmonary disease, renal failure, major liver dysfunction within the last 2 years, digestive disorders including gastric reflux, irritable bowel disease, Crohn's disease or related conditions current smoker or recently quit less than 6 months prior) or medications that would prevent the ability to comply with treatment assignment (e.g. blood thinners, arrhythmia control medications, prescription narcotic pain medications).
* Use of estrogen or testosterone replacement therapy within the past 6 months,
* Current use of oral corticosteroids > 5 days/month on average
* Cold, flu, virus, allergy or other conditions that impairs sensory perceptions (taste and smell) which may impact protocol compliance
* COVID19 positive status at time of enrollment
* Consumes an average of ≥1 serving of turmeric per day, or has never consumed and/or would not be willing to consume turmeric
* Consumes black pepper ≥ 3 servings per day and/or would not be willing to abstain from pepper consumption for the prescribed days during the study
* Abstinence from or dislike of either turmeric or black pepper
* Dependence on others for food procurement and preparation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 7 days
  Self-reported pain according to Numeric Rating Scale (NRS), score from 0 = no pain, 10 = worst pain, within each 7-day intervention (placebo, turmeric, turmeric+black pepper)

SECONDARY OUTCOMES:
Physical Activity | 7 days
  Minutes of physical activity per week at moderate and vigorous intensity physical activity levels, and minutes of sedentary behavior, assessed via accelerometry
Pain Survey | Once per week during the 3 week (21-day) study
Insulin | Baseline and every 7 days during the 21-day study
  (uU/ml)
C-reactive protein | Baseline and every 7 days during the 21-day study
  (ug/ml)
IL-6 | Baseline and every 7 days during the 21-day study
  Interleukin 6 (pg/ml)
IL-10 | Baseline and every 7 days during the 21-day study
  Interleukin 10 (pg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data (including data dictionaries) will be shared or made publicly available for any publication of findings.
Time Frame: Immediately following publication.
Access Criteria: Public repository